CLINICAL TRIAL: NCT02876419
Title: A Long Term Follow-up Study of Patients From the REP 301 Protocol
Status: Completed | Type: Observational
Sponsor: Replicor Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: REP 301-LTF
Record Dates: First submitted 2016-08-16; First posted 2016-08-23 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis B, Chronic; Hepatitis D, Chronic
Keywords: nucleic acid polymer REP 2139 HBsAg hepatitis B hepatitis D
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis D, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Frozen serum containing viral DNA / RNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The REP 301 treatment protocol involved the treatment of patients with chronic hepatitis B / hepatitis D co-infection with two agents: REP 2139-Ca and pegylated interferon (peg-IFN). In this protocol, similar reduction/clearance of serum HBsAg and improved response to immunotherapy were observed in addition to clearance of serum HDV RNA. The REP 301 protocol was designed to include a 24 week follow-up period after treatment, however given the strong antiviral response against HBV and HDV infection in these patients, it is now important to extend the follow-up period in these patients to monitor over a longer period after treatment the safety and efficacy combined REP 2139-Ca / peg-IFN treatment in patients in the REP 301 protocol.

DETAILED DESCRIPTION:
The REP 301-LTF is a long-term follow-up, non-blinded study of patients from the REP 301 protocol. In this study, all eligible patients from the REP 301 protocol will have their followup evaluation extended for an additional 3 years, consisting of 6 visits scheduled every 6 months following the last follow-up visit scheduled in the REP 301 protocol. During each visit a physical examination and documentation of any symptoms, experiences will be conducted as well as blood tests for safety and virology as described below. This study will examine the long term safety effects in patients who have completed of treatment exposure in the REP 301 trial (REP 2139-Ca therapy for 30 weeks and PEG-IFN taken for 48 weeks with a 15 week overlap in combination) and the duration of suppression of serum HBV and HDV viremia observed in the REP 301 protocol. This requires that subjects have completed antiviral treatment in the REP 301 protocol and are not immediately transitioned to further antiviral treatment unless necessary. The total duration of this study for each subject is 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.

Exclusion Criteria:

1. Any patients not enrolled in the REP 301 protocol or not successfully completing all treatment and follow-up visits in the REP 301 protocol
2. A history of alcohol abuse within the last year
3. The use of illicit drugs within the past two years.
4. Inability to provide informed consent.
5. Inability or unwillingness to provide blood samples.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients completing treatment exposure in the REP 301 protocol.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-08; Primary Completion 2019-11-13 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Long term safety (test abnormalities) | 3 years
  The proportion of patients with emergent lab test abnormalities.
Long term safety (AEs) | 3 years
  Proportion of patients with adverse events.
Long term safety (SAEs) | 3 years
  Proportion of patients with serious adverse events.

SECONDARY OUTCOMES:
Long term efficacy (serum HBsAg) | 3 years
  Proportion of patients who maintain serum HBsAg < 1 IU/ml.
Long term efficacy (serum anti-HBs) | 3 years
  Proportion of subjects who maintain anti-HBs titers above 10 mIU/ml.
Long term efficacy (serum HBV DNA) | 3 years
  Proportion of patients who maintain serum HBV DNA < 10 IU / ml.
Long term efficacy (serum HDV RNA) | 3 years
  Proportion of patients who maintain undetectable serum HDV RNA (target not detected).

CONTACTS AND LOCATIONS:
Overall Officials: Victor Pantea, MD, Principal Investigator — Infectious Clinical Hospital (n.a. Toma Ciorba)
Locations (1):
- Infectious Clinical Hospital (n.a. Toma Ciorba), Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bazinet M, Pantea V, Cebotarescu V, Cojuhari L, Jimbei P, Anderson M, Gersch J, Holzmayer V, Elsner C, Krawczyk A, Kuhns MC, Cloherty G, Dittmer U, Vaillant A. Persistent Control of Hepatitis B Virus and Hepatitis Delta Virus Infection Following REP 2139-Ca and Pegylated Interferon Therapy in Chronic Hepatitis B Virus/Hepatitis Delta Virus Coinfection. Hepatol Commun. 2020 Nov 13;5(2):189-202. doi: 10.1002/hep4.1633. eCollection 2021 Feb. PMID 33553968
- [Derived] Bazinet M, Pantea V, Cebotarescu V, Cojuhari L, Jimbei P, Albrecht J, Schmid P, Le Gal F, Gordien E, Krawczyk A, Mijocevic H, Karimzadeh H, Roggendorf M, Vaillant A. Safety and efficacy of REP 2139 and pegylated interferon alfa-2a for treatment-naive patients with chronic hepatitis B virus and hepatitis D virus co-infection (REP 301 and REP 301-LTF): a non-randomised, open-label, phase 2 trial. Lancet Gastroenterol Hepatol. 2017 Dec;2(12):877-889. doi: 10.1016/S2468-1253(17)30288-1. Epub 2017 Sep 28. PMID 28964701